CLINICAL TRIAL: NCT00335946
Title: A Pilot Investigational Study: Treatment of Anxiety With Non-Needle Electro-Acupuncture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0602060019
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-07

CONDITIONS: Anxiety, Mild to Moderate
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HANS non-needle acupuncture
Procedure: Stimulation of two acupuncture points bi-lateral

SUMMARY:
The purpose of this study is to determine the effects of non-needle electro-acupuncture on mild to moderate anxiety. The hypothesis is that this style of treatment will reduce state anxiety and not trait anxiety as measured by the Spielberger STAI test.

DETAILED DESCRIPTION:
Persistent and unrelenting stress is defined as anxiety. Anxiety disorders are among the most common mental disorders in society. The NIH estimates that nearly 200 million Americans suffer from anxiety. Anxiety disorders are associated with a lower quality of life, functional impairment and disability, and are also associated with co-morbid physical illness.

Acupuncture, one form of complementary and alternative medicine, has been used to treat anxiety. Non-needle acupuncture is one of the safest methods, with none to rare side effects. This method has been studied in China (Han 1986) and America (Ulett 1998) Pre-intervention testing, then three treatments within one week, will be followed by post intervention testing.

ELIGIBILITY:
Inclusion Criteria: Normally healthy persons with mild to moderate anxiety -

Exclusion Criteria: Severe anxiety, depression, pregnancy, and previous experience with HANS non-needle electro-acupuncture treatment

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Spielberger STAI test

CONTACTS AND LOCATIONS:
Overall Officials: David V. Beavers, DC, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chirpractic, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Ulett GA, Han J, Han S. Traditional and evidence-based acupuncture: history, mechanisms, and present status. South Med J. 1998 Dec;91(12):1115-20. doi: 10.1097/00007611-199812000-00004. PMID 9853722
- [Background] Zhang H, Zeng Z, Deng H. Acupuncture treatment for 157 cases of anxiety neurosis. J Tradit Chin Med. 2003 Mar;23(1):55-6. No abstract available. PMID 12747204
- [Background] Han JS. Electroacupuncture: an alternative to antidepressants for treating affective diseases? Int J Neurosci. 1986 Mar;29(1-2):79-92. doi: 10.3109/00207458608985638. PMID 3516903
- [Background] Jorm AF, Christensen H, Griffiths KM, Parslow RA, Rodgers B, Blewitt KA. Effectiveness of complementary and self-help treatments for anxiety disorders. Med J Aust. 2004 Oct 4;181(S7):S29-46. doi: 10.5694/j.1326-5377.2004.tb06352.x. PMID 15462640
- [Background] Mamtani R, Cimino A. A primer of complementary and alternative medicine and its relevance in the treatment of mental health problems. Psychiatr Q. 2002 Winter;73(4):367-81. doi: 10.1023/a:1020472218839. PMID 12418362
- [Background] Tang J, Gibson SJ. A psychophysical evaluation of the relationship between trait anxiety, pain perception, and induced state anxiety. J Pain. 2005 Sep;6(9):612-9. doi: 10.1016/j.jpain.2005.03.009. PMID 16139780